CLINICAL TRIAL: NCT05910216
Title: Online Dance Versus Online Therapeutic Exercise on Quality of Life - A Protocol for a Randomized Controlled Trial Investigating Social Telerehabilitation Efficacy in Parkinson's Disease.
Brief Title: Online Dance Versus Therapeutic Exercise for Parkinson Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONLINEREHABPD
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Dance; Physiotherapy; Telehealth; Telerehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Dance & Music (Online) (Experimental): Social Telerehabilitation with Dance & Music (Online): The dance intervention will be instructed by a physiotherapist and dance professional, who will follow a structure based on the materials of the Dance for Parkinson's (USA) ® method
  Interventions: Other: Dance & Music (Online)
- Group Multimodal Therapeutic Exercise & Music (Online) (Active Comparator): Social Telerehabilitation with Multimodal Therapeutic Exercise & Music (Online): The intervention with multimodal therapeutic exercise will be instructed by a physiotherapist, who will follow a structure based on a previous study and Physical Therapy Guidelines for People with PD
  Interventions: Other: Multimodal Therapeutic Exercise & Music (Online)

INTERVENTIONS:
Other: Dance & Music (Online) — This is a social telerehabilitation with dance and music. It will include artistic form, imageries using scenic arts, imageries using aspects of theater and storytelling, movement improvisation, choreography and sequence of movements, complex dance movements, fluidity of movement or connection between one movement and another, rhythmicity and/or movement built with music. It will include instructions for motor learning, music, and socialization
  Arms: Group Dance & Music (Online)
Other: Multimodal Therapeutic Exercise & Music (Online) — This is a social telerehabilitation with multimodal therapeutic Exercise and Music. It is restricted to the execution of movements within series and standardized and fixed repetitions, with a background music. It will not include dance. It will include instructions for motor learning, music, and socialization.
  Arms: Group Multimodal Therapeutic Exercise & Music (Online)

SUMMARY:
This is a randomized clinical trial in an online format, which will only include people with PD randomly divided into two groups:

Group 1 - Social Telerehabilitation with Dance and Music Group 2 - Social Telerehabilitation with Multimodal Therapeutic Exercise and Music

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic PD according to the clinical criteria of the London Brain Bank Criteria (2006);
* Age between 40-90 years;
* A minimum score of 18 in the Montreal Cognitive Assessment;
* Drug therapy/exercise stable for at least four weeks before the study starts;
* Agreement to participate in the study according to the Informed Consent Form.

Exclusion Criteria:

* Auditory and/or visual disturbances that compromise understanding simple commands;
* Access to the internet and a device to access online classes;
* A house member and/or caregiver at home for supervision during the entire experiment, including evaluations and interventions. For patients scoring less than 2.5 points on the modified Hoehn and Yahr Scale (indicating mild disease impairment, independence in daily living activities, and no risk of falls), the requirement for household member supervision may be waived.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Quality of life | Change from Pre to Post treatment (12 weeks) and FOLLOW-UP (after 4 weeks of study ending)
  Quality of life measured by Parkinson's Disease Questionnaire (PDQ-39). Scores range from 0-100 (100 = maximum level of problems).
Assessment of Well-being | Change from Pre to Post treatment (12 weeks) and FOLLOW-UP (after 4 weeks of study ending)
  Well-being measured by the scale Positive and Negative Affect Scale (PANAS). scores range from 10 - 50, a higher score indicates more of a positive affect.

SECONDARY OUTCOMES:
Assessment of Motor symptoms severity | Change from Pre to Post treatment (12 weeks) and FOLLOW-UP (after 4 weeks of study ending)
  Motor symptoms severity measured by the scale Unified Parkinson's disease rating scale, motor subscale (UPDRS III). Part III: Motor examination: 18 items. Score range: 0-132, 32 and below is mild, 59 and above is severe.
Assessment of Functional lower extremity strength | Change from Pre to Post treatment (12 weeks)
  Functional lower extremity strength measured by the Five times sit to stand test (FTSTS). The time to complete the test is measured, where lower time to perform sit to stand represents better functional lower extremity strength
Assessment of Symptoms of Anxiety | Change from Pre to Post treatment (12 weeks)
  Symptoms of Anxiety measured by the Parkinson Anxiety Scale (PAS). Scores range from 0-48 (48= maximum level of problems).
Assessment of Attention and Memory Recognition | Change from Pre to Post treatment (12 weeks)
  Executive function by means attention and memory recognition measureb by Online Attention Test (OAT) and Recognition Memory Test (RMT).
Feasibility (self-perceptions) | Change from Pre to Post treatment (12 weeks)
  Self-perceptions (feasibility) of technology usability, socialization and benefits of interventions based on a structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Pagnussat, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Aline, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided